CLINICAL TRIAL: NCT00411034
Title: A Repeated-Dose Evaluation of Analgesic Use and Safety of Dilaudid SR( Hydromorphone HCI) in Patients With Chronic Cancer Pain
Brief Title: A Repeated-Dose Evaluation of Use of a Pain Relieving Drug and Safety of OROS Hydromorphone HCI in Patients With Chronic Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011614
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Analgesics, Opioid; Pain
Keywords: Opioids; Chronic Cancer Pain; analgesic
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: OROS Hydromorphone HCI

SUMMARY:
The purpose of this repeated dose study is to develop recommended dosing information for initiation of therapy with OROS Hydromorphone HCI (slow release) in patients with chronic cancer pain converting from other strong oral or transdermal opioids. It will also assist in the development of a recommended starting dose by which patients can be titrated to an appropriate maintenance dose of OROS hydromorphone HCI (slow release). The safety profile for OROS Hydromorphone HCI (slow release) will also be evaluated.

DETAILED DESCRIPTION:
This randomized (patients assigned to treatment by chance), single-blind (with respect to dose), open-label (patients know what study treatment, not dose, they are receiving) repeated dose study evaluating patients with chronic cancer pain was conducted in tandem (together) with a similar protocol in patients with chronic non-malignant pain. A total of 463 patients were enrolled and evaluated in these studies. Patients receiving chronic opioid therapy were converted to once daily OROS hydromorphone (slow release) using oral morphine equivalents. Supplementary immediate-release (IR) hydromorphone was provided for breakthrough pain. The dose of OROS hydromorphone (slow release) was escalated after every 2 days of therapy until no more than 3 doses of immediate-release (IR) hydromorphone were required in a 24-hour period. Once a patient could be maintained on a stable dose of OROS hydromorphone (slow release) for 3 consecutive days, the patient entered a 2-week maintenance phase. Patients who completed the study were eligible for participation in an OROS hydromorphone (slow release) long-term extension study, Study DO-109. The hypothesis is the 24-hour controlled-release form of oral hydromorphone may provide consistent pain relief, convenient dosing, and enhanced compliance while possibly decreasing the incidence of side effects associated with peak (high) and trough (low) fluctuations in plasma drug concentrations typically seen with immediate-release dosage formulations. Patients received OROS Hydromorphone HCI (slow release) at Visit 2,3, and 4 (either 8,16,32, and/or 64mg tablets) taken orally. OROS Hydromorphone HCI (slow release) doses were titrated after every two days of therapy as necessary until dose stabilization occured, followed by a two week Maintenance Therapy Phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic cancer pain who are currently receiving strong oral or transdermal opioid analgesics or patients suitable for advancement of therapy to step 3 on the WHO (World Health Organization) analgesic ladder
* patients who can reasonably be expected to have stable opioid requirements for the duration of the study

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone (or other opioid agonists)
* patients who are pregnant or breast-feeding
* patients with severe respiratory compromise or severely depressed ventilatory function
* patients with any gastrointestinal disorder or acute abdominal conditions including pre-existing severe GI narrowing (pathologic or iatrogenic), that may affect the absorption or transit of orally administered drugs
* patients with clinically significant impaired renal or hepatic function, Addison's disease, hypothyroidism, prostatic hypertrophy, or urethral stricture, dysphagia or are unable to swallow tablets or any significant CNS disorder, including but not limited to head injury, intracranial lesion, increased intracranial pressure, seizure disorder, stroke within the past 6 months, and disorders of cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
No primary efficacy variable was defined in report. Protocol variables measured included: Total daily dose of OROS hydromorphone, daily use of rescue medication, daily pain relief scores, and time/number of steps needed for dose stabilization.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA